CLINICAL TRIAL: NCT02254759
Title: A Study of RO5186582 Treatment on Cytochrome P450 (CYP) 3A4 Activity in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: WP29393; 2014-001850-41 (EudraCT Number)
Record Dates: First submitted 2014-09-23; First posted 2014-10-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Midazolam

ARMS (5):
- IV Midazolam Alone (Other): A single 1 milligram (mg) dose of IV Midazolam on Day 1.
  Interventions: Drug: Midazolam, IV
- Oral Midazolam Alone (Other): A single 5 mg oral dose of midazolam on Day 2.
  Interventions: Drug: Midazolam, oral
- RO5186582 Alone (Experimental): RO5186582 240 mg oral tablet twice daily (BID) for 14 days from Days 3 to 16.
  Interventions: Drug: RO5186582
- RO5186582 Plus IV Midazolam (Experimental): RO5186582 240 mg BID oral tablet in combination with a single 1 mg IV dose of midazolam on Day 17.
  Interventions: Drug: Midazolam, IV; Drug: RO5186582
- RO5186582 Plus Oral Midazolam (Experimental): RO5186582 240 mg BID in combination with a single 5 mg oral dose of midazolam on Day 18.
  Interventions: Drug: Midazolam, oral; Drug: RO5186582

INTERVENTIONS:
Drug: Midazolam, IV — 2 milligrams per milliliter (mg/mL) midazolam solution for IV administration. For a 1 mg dose, the midazolam solution (0.5 mL of 2 mg/mL) will be injected at 2 milligrams per minute (mg/min).
  Arms: IV Midazolam Alone; RO5186582 Plus IV Midazolam
Drug: Midazolam, oral — 0.1 mg/mL midazolam for oral administration. For a 5 mg dose, participants will receive 50 mL of 0.1 mg/mL midazolam.
  Arms: Oral Midazolam Alone; RO5186582 Plus Oral Midazolam
Drug: RO5186582 — RO5186582 120 mg film-coated release tablet.
  Arms: RO5186582 Alone; RO5186582 Plus IV Midazolam; RO5186582 Plus Oral Midazolam

SUMMARY:
This is a non-randomized, open-label, five treatment, fixed sequence cross-over study to investigate the effect of RO5186582 treatment on CYP3A activity using midazolam as a probe CYP3A substrate, and also to assess the pharmacodynamic measures of brain electrical activity and sedation to explore the pharmacodynamic interaction between the gama-amino butyric acid (GABA)A negative allosteric modulator RO5186582 and the prototypical GABAA positive allosteric modulator midazolam. The anticipated study duration is up to nine weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants with signed informed consent.

Exclusion Criteria:

* A history of epilepsy, convulsions or significant head injury
* Significant history of drug allergy, as determined by the Investigator, or a known hypersensitivity to any of the ingredients of any of the study treatments
* Use of any drugs or substances, including herbal treatments such as St John's Wort, that are known to be substrates, inducers or inhibitors of CYP3A4 within 30 days of the first dose administration
* Pregnant or lactating
* Any other clinically relevant abnormalities, concomitant diseases or ongoing medical conditions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Bioavailability of Drug (F) for Oral Midazolam | Pre-dose [-0.5 hour (h)] and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10 and 14 h post-dose (pd) on Day (D) 2 and 18, and 22 h pd on D3 and 19
Total Plasma Clearence (CL) for IV Midazolam | Pre-dose [-10 minutes (min)] and 0.08 (5 min), 0.25 (15 min), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 14 h pd on D1 and D17, and 22 h pd on D2 and D18
Apparent Volume of Distribution at Steady-State (Vss) for IV Midazolam | Pre-dose (-10 min) and 0.08 (5 min), 0.25 (15 min), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 14 h pd on D1 and D17, and 22 h pd on D2 and D18
Maximum Observed Plasma Concentration (Cmax) for Oral Midazolam | Pre-dose (-0.5 h) and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10 and 14 h pd on D2 and 18, and 22 h pd on D3 and D19

SECONDARY OUTCOMES:
Apparent Volume of Distribution (V/F) for Oral Midazolam | Pre-dose (-0.5 h) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 14 h pd on D2 and D18, and 22 h pd on D3 and D19
Area Under the Plasma Concentration Time Curve from Time Zero to Time Tau, Where Tau is the Dosing Interval (AUC0-tau) for RO5186582 and RO5271857 (metabolite of RO5186582) | D18: Pre-dose -0.17 h (10 min) and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10 and 12 h pd
Cmax for RO5186582 and RO5271857 (metabolite of RO5186582) | Pre-dose (10 min) and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10 and 12 h pd on D18 (timepoints relative to oral midazolam dosing are (- 2 h 10 min), -1.5, -1, -0.5, 0 h pre-dose and 1, 2, 3, 4, 6, 8, and 10 h pd)
Tmax for RO5186582 and RO5271857 (metabolite of RO5186582) | Pre-dose (10 min) and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10 and 12 h pd on D18 (timepoints relative to oral midazolam dosing are (- 2 h 10 min), -1.5, -1, -0.5, 0 h pre-dose and 1, 2, 3, 4, 6, 8, and 10 h pd)
Metabolic Ratio Based on AUC0-inf for IV Midazolam | Pre-dose (-10 min) and 0.08 (5 min), 0.25 (15 min), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 14 h pd on D1 and D17, and 22 h pd on D2 and D18
Change From Baseline in Event-Related Potential (ERP) parameters Using Oddball Auditory | D-1 (Baseline) and D16 at 1 and 4 h pd, time-matched to planned time, and D2 and D8 at 1 and 4 h pd
Change from Baseline in Electroencephalogram (EEG) Parameters | D-1 (Baseline) and D16 at 1 and 4 h pd, time-matched to planned time, and D2 and D8 at 1 and 4 h pd
Change From Baseline in Saccadic Eye Movement (SEM) Parameters | D-1 (Baseline) and D16 at 1 h pd, time-matched to planned time, and D2 and D18 at 1 h pd
Change From Baseline in Attention and Memory of Selected Domains of Repeatable Battery for the Assessment of Neuropyschological Status (RBANSTM) | D-1 (Baseline) and D16 at 2 and 5 h pd, time-matched to planned time, and D2 and D18 at 2 and 5 h pd
Change from Baseline in Concentration of 4 Beta-Hydroxy Cholesterol | D1 (Baseline) and D17
Area Under the Plasma Concentration Time Curve from Zero to Infinity (AUC0-inf) for Oral and IV Midazolam | Midazolam (MDZ)-oral: pre-dose (-0.5 h) and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10 and 14 h pd on D2 and 18, and 22 h pd on D3 and 19; MDZ-IV: Pre-dose (-10 min) and 5, 15 min, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 14 h pd on D1 and 17, and 22 h pd on D2 and 18
Cmax for IV Midazolam | Pre-dose (-10 min) and 5, 15 min, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 14 h pd on D1 and 17, and 22 h pd on D2 and 18
Area Under the Plasma Concentration Time Curve from Zero to Last Measurable Concentration (AUC[0-last]) for Oral and IV Midazolam | MDZ-oral: pre-dose (-0.5 h) and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10 and 14 h pd on D2 and 18, and 22 h pd on D3 and 19; MDZ-IV: Pre-dose (-10 min) and 5, 15 min, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 14 h pd on D1 and 17, and 22 h pd on D2 and 18
Time to Maximum Observed Concentration (Tmax) for Oral and IV Midazolam | MDZ-oral: pre-dose (-0.5 h) and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10 and 14 h pd on D2 and 18, and 22 h pd on D3 and 19; MDZ-IV: Pre-dose (-10 min) and 5, 15 min, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 14 h pd on D1 and 17, and 22 h pd on D2 and 18
Terminal Elimination Half-Life (t1/2) for Oral and IV Midazolam | MDZ-oral: pre-dose (-0.5 h) and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10 and 14 h pd on D2 and 18, and 22 h pd on D3 and 19; MDZ-IV: Pre-dose (-10 min) and 5, 15 min, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 14 h pd on D1 and 17, and 22 h pd on D2 and 18
Apparent Clearence (CL/F) for Oral Midazolam | Pre-dose (-0.5 h) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 14 h pd on D2 and D18, and 22 h pd on D3 and D19

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Leeds, United Kingdom